CLINICAL TRIAL: NCT02138864
Title: Targeting Monoaminergic Neuronal Networks in the Parkinsonian Patients After Carbon Monoxide Intoxication
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, chiungchihchang, MD, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 101-4350A; CDE102IND01009 (Registry Identifier: CHIUNH-CHIH CHANG)
Record Dates: First submitted 2014-05-07; First posted 2014-05-15 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Carbon Monoxide-induced Parkinsonism
Keywords: carbon monoxide intoxication; Parkinsonism; 18F-DTBZ AV-133
MeSH Terms: conditions — Carbon Monoxide Poisoning; Parkinsonian Disorders | interventions — florbenazine F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-FP-(+)-DTBZ only (Experimental): PET tracer: 18F-FP-(+)-DTBZ
  Interventions: Radiation: 18F-FP-(+)-DTBZ

INTERVENTIONS:
Radiation: 18F-FP-(+)-DTBZ — no available

SUMMARY:
The study purpose is to determine the clinical values of 18F-FP-(+)-DTBZ in the diagnosis of Parkinsonism in patients with carbon monoxide intoxication, regional distribution and its correlation with clinical parameters. This study is expected to be completed in a period of 3 years.

DETAILED DESCRIPTION:
With the urbanization of Taiwanese society, there are increasing numbers of people committing suicide by charcoal burning, making carbon monoxide (CO) encephalopathy a new pandemic phenomenon. In CO related parkinsonism, the clinical features included gait disturbances, mask face, rigidities and small steps. From literature searches, the CO related parkinsonism is related to white matter damages or decline in dopamine innervations. From our previous research results, the CO related neuronal damages would started from reversible or progressive white matter demyelination. For some patients, axonopathy or gray matter atrophy developed and became irreversible. The neuronal networks in determining development of Parkinsonism required to be established.

In terms of neurotransmitter, most of the clinical data for Parkinsonism came from studies of idiopathic Parkinson's disease while the data of CO related Parkinsonism were limited to case reports. From neuropathology studies in idiopathic Parkinson's disease, dopamine deficits and decreased in monoamine transporters were observed well before the development of clinical features. Although there is linkage between CO related Parkinsonism and dopamine deficits, patients with CO intoxication had poor response to levodopa. The observation suggested the critical networks and neurotransmitters were still not well understood.

18F-FP-(+)-DTBZ is a newly developed nuclear medicine tracer for monoamine transporter. The study purpose is to determine the clinical values of 18F-FP-(+)-DTBZ in the diagnosis of Parkinsonism in patients with carbon monoxide intoxication, regional distribution and its correlation with clinical parameters. This is a three-year prospective research. For each patient, the PET will be arranged twice, with an interval of 18 months. The regional distribuation of 18F-FP-(+)-DTBZ in relation to Parkinsonism severity and regional reduction patterns longitudially will be assessed in order to understand the regional neurotoxicity and the functional progression.

ELIGIBILITY:
Inclusion criteria

1. Male or female age 20 years to 65 years.
2. Patients group should fulfilled diagnostic criteria of carbon monoxide intoxication
3. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm consent)

Exclusion criteria

1. History of developmental disorders, agitated mood or a confused state that prevented either a neuropsychiatric interview or neuroimaging.
2. Unable to stay still in the PET scanner for 30 minutes.
3. History or presence of QTc prolongation. (>500msec)
4. Pregnancy and breast feeding.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Assess the regional decline in 18F-DTBZ uptake of Parkinsonism after carbon monoxide intoxication | up to 3 years
  This study will assess the brain uptake and distribution of 18F-DTBZ in 25 carbon monoxide intoxication patients with Parkinsonism. For each patient, the PET will be arranged twice, with an interval of 1.5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Chiung-Chih Chang, M.D.; Ph.D, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan